CLINICAL TRIAL: NCT05605444
Title: The Effect of an Acute Bout of Exercise on Pain Sensitivity and Clinical Pain in Adults With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taif University (Other)
Responsible Party: Principal Investigator, Hosam Alzahrani, Assistant Professor, Taif University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-02-K-076-0722-770
Record Dates: First submitted 2022-10-16; First posted 2022-11-04 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Osteoarthritis, Knee
Keywords: acute bout of exercise; Pain sensitivity; Clinical pain
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Isometric exercise-one repetition (Experimental): Isometric exercise consisting of 1 session only. The session will last for around 5 minutes which will include asking the patient to do 1 repetition of wall squat for 3 min or to volitional fatigue at 100° knee angle.
  Interventions: Other: Single bout of exercise
- Isometric exercise-three repetitions (Experimental): Isometric exercise consisting of 1 session only. The session will last for around 10 minutes which will include asking the patient to perform 3 repetition of wall squat (each time the exercise will be performed for 3 min or to volitional fatigue at 100°degree knee angle); patient will be given 30 sec rest between repetitions.
  Interventions: Other: Single bout of exercise
- Control (no intervention) (No Intervention): Will not receive any intervention

INTERVENTIONS:
Other: Single bout of exercise — isometric wall squat at a knee joint angle of 100 degrees. Instruct participant to place their back against the wall with feet positioned parallel and spaced shoulder-width apart. Lower themselves down until they reached a knee joint angle of 100 degrees. Measure knee joint angle by placing a goniometer on the lateral epicondyle of the knee, in line with the femur whilst the anchor arm was in line with the lateral malleolus.
  Arms: Isometric exercise-one repetition; Isometric exercise-three repetitions

SUMMARY:
The goal of this interventional study is to investigate the effectiveness of an acute bout of exercises on pain sensitivity and clinical pain among adults with knee osteoarthritis. The following question will be answered in this research Q1: Is acute bout of exercise effective in reducing pain sensitivity and intensity among adult with knee osteoarthritis?

Participants who agree to participate and sign the informed consent will be randomised to one of three groups:

Group 1: Isometric exercise with neutral language and no verbal suggestion consisting of 1 rep of wall squat, 3 min or to volitional fatigue at 100° knee angle;(n=30).

Group 2: Isometric exercise with neutral language and no verbal suggestion consisting of 3 reps of wall squat, 3 min or to volitional fatigue at 100°degree knee angle, 30 sec rest between rep, ;(n=30).

Group 3 (Control group): true control (do nothing);(n=30).

DETAILED DESCRIPTION:
Osteoarthritis (OA) has been defined as losing the function of cartilage which causes inflammation and pain. OA is one of the most common joint diseases affecting both men and women worldwide, with women being more affected than men. A previous report estimated that that OA affects approximately 240 million people globally. Furthermore, the 2016 Global Burden of Disease Study estimated that the global incidence of hip and knee OA is 199 cases per 100,000, with incidence rates varying by region and ethnicity. The economic impact of osteoarthritis is significant, and it continues to increase as the population ages and obesity increases.

The knee OA has more clinical symptoms than any other form of OA. Knee OA results not only in pain, but also causes loss of function, and decreased quality of life. The typical clinical presentation of Knee OA is knee pain, brief morning stiffness (less than 30 minutes), crepitus, bony tenderness, and enlargement without palpable warmth, muscles weakness. Furthermore, people diagnosed with OA commonly report psychological problems such as anxiety and fear of movement. These problems might prevent people from participation in exercise and social events, leading to further physical and social isolation. The prevalence of knee OA is estimated to be about 33% and it is one of the five causes of disability among people, especially in the elderly individuals.

Alleviating pain is critical to improve the lives of people with Knee OA. Exercise training is a fundamental treatment modality for chronic low back pain, knee osteoarthritis OA and fibromyalgia. However, pain intensity, kinesiophobia and low self-efficacy are barriers to initiating and adhering to an exercise training program. Therefore, an effective strategy to reduce pain intensity, kinesiophobia and increase self-efficacy to facilitate participation in an exercise training program for people with chronic musculoskeletal pain conditions is important. A single acute bout of exercise can produce a consistent reduction in pain sensitivity, termed exercise induced hypoalgesia, in pain-free populations. Although, the hypoalgesia response is likely dependent on the exercise mode or prescription variables applied. In chronic pain populations, exercise induced hypoalgesia is not always consistent, the optimal exercise dose is largely unknown and there are few studies in people with chronic low back pain, fibromyalgia and knee OA. It is not clear whether a single bout of exercise results in a clinically meaningful reduction in pain sensitivity or clinical pain intensity in these population groups. Pilot data from our lab showed adults with chronic low back pain (n=21) reduced pain sensitivity (via pain pressure threshold) globally (Cohen's d=0.5; medium effect), local to the site of pain (low back; d=0.5; medium effect) and distal to the site of pain (leg; d=0.8; large effect) following a single wall squat (100° knee angle) for three minutes or until volitional fatigue. Given these promising results, exploring the utility of this approach in a controlled clinical setting across a range of common chronic pain conditions is warranted to establish efficacy.

Methods Ethics The trial protocol was approved for the study protocol by the General Administration for Research and Studies of the Directorate of Health Affairs, Makkah, Saudi Arabia (H-02-K-076-0722-770). This study will follow the Declarations of Helsinki. Consents will be obtained from the patients before participating in the study.

Study design:

This study design will be a randomized controlled trial with a pre-post control design.

Settings:

The trial will be performed at the Department of Physiotherapy at King Abdul-Aziz Hospital and King Faisal Hospital in Makkah in Saudi Arabia.

Sample size:

Based on sample size calculation following pilot study conducted in our lab, we plan to enroll 90 participants in the study with symptomatic knee osteoarthritis. Participants will be randomly divided into three groups. Each group contains 30 individuals. The aim is to achieve 90% power to observe a significant difference of 5% (alpha of 0.05) using a two-tailed t-test.

Sampling techniques:

Participants will be recruited using consecutive sampling technique. Simple randomization will be used to allocate participants in each group. Participants will be stratified based on sex and then allocated to each group in a 1:1 ratio. Randomization will be conducted by a participant who is not involved in the study.

Data analysis:

Data analysis will be performed using R software (version 4.2.0; R Foundation for Statistical Computing, Vienna, Austria). Baseline characteristics will be summarized using descriptive statistics; continuous variables will be expressed as the mean and standard deviations, while categorical variables will be reported as frequencies and percentages. Separate linear mixed-effects models will be constructed to examine the effects of interventions over time, utilizing the "lme4" package for model fitting and the "lmerTest" package to facilitate hypothesis testing, including calculations of p-values and 95% confidence intervals. The "emmeans" package will be employed for post hoc analyses, specifically for estimating marginal means and performing comparisons between group levels.

For the within-group analyses, separate LMMs will be developed for each intervention group. These models will include random and fixed effects for time to capture within-group changes over time for each outcome.

Between-group differences over time will be analyzed using LMMs that will incorporate fixed effects for time, group, and a time-by-group interaction term. This approach will aim to identify differential responses to exercise interventions across groups. Random intercepts will be incorporated into all models to account for the inherent correlation of repeated measures within the subjects.

All models will be estimated using restricted maximum likelihood to ensure unbiased variance component estimates, particularly when comparing models with different fixed effects structures. The analysis will adopt an intention-to-treat approach to analyze participants according to their original group assignments. A significance level of 0.05 will be used for all inferential statistics.

An exploratory analysis will be conducted to investigate the differences between the two intervention groups for squat hold time under tension, and across the three groups for expectations of changes in PPT and knee pain intensity. Owing to the violations of normality assumptions for both the squat-hold total time under tension and the expected data, non-parametric analyses using the Mann-Whitney U test and Kruskal-Wallis test will be employed to compare squat-hold total time under tension and self-reported expectations, respectively, between groups.

Additionally, post-hoc analyses will be performed using LMM to determine whether there will be a three-way interaction effect between the total squat hold time under tension, group, and time on the PPT and VAS. This approach will allow us to account for within-subject variability by including random intercepts for participants.

Safety and adverse events:

Exercise programs are generally safe; however, it is possible that participants may experience some unforeseen problems such as muscle soreness, falls or other injuries. Participants will be closely monitored to keep track of any unwanted effects or any problems. If there are any unwanted effects the program may be stopped and the reasons will be discussed with the treating physiotherapist and investigator. In case of a serious adverse event, participants will be advised to seek immediate medical assistance.

Funding:

We will apply for funding from Taif University.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older.
2. Diagnosed by surgeon using radiological imaging and clinical decision with unilateral or bilateral symptomatic knee OA.
3. Have chronic knee pain for three months and more (with average VAS in the last week >= 3/10).
4. Able to perform physical therapy exercise.

Exclusion Criteria:

1. Pregnancy.
2. Severe musculoskeletal or neuromuscular disorders or any disease that prevent performing exercises.
3. Uncontrolled diabetes.
4. Knee or lower limb surgery.
5. Sensations problems.
6. Orthopedic impairment (e.g., sever deformities, ligament injuries, balance problems and fractures in lower limb in the last 6 months).
7. Any contraindication to exercise preventing them from performing exercises as per the "American College of Sports Medicine" guidelines.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Pain pressure threshold | Change from pre-intervention (baseline) compared to post-intervention (immediately after session)
  The pain will be measured using digital pressure algometer, FDX®️ (Wagner instrument, Greenwich, USA). All trials will be conducted on forearm, lumbar spine and calf sites. There will be at least 20 sec rest before an individual site is tested again. Two trials will be performed at each site. The raw values of each test will be recorded.
  Because we are testing repeated times, we will use a marker to mark the location of each test site to ensure consistency in location.
  Algometer must be positioned perpendicular to the measurement site for all trials.

SECONDARY OUTCOMES:
Pain intensity | Change from pre-intervention (baseline) compared to post-intervention (immediately after session)
  It will be measured using Visual Analogue Scale (VAS; 0-10). A rating of zero means that participant don't currently have pain at the low back. A rating of ten on this scale means that the pain at low back is the worst pain. So, the higher the number on this scale means the higher the pain intensity participant is experiencing.

CONTACTS AND LOCATIONS:
Overall Officials: Hosam Alzahrani, PhD, Principal Investigator — Taif University, College of Applied Medical Science, Physical Therapy Department, TAIF, SAUDI ARABIA
Locations (1):
- King AbdulAziz Hospital and King Faisal Hospital, Mecca, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Zabarmawi J, Miller CT, Owen PJ, Mundell NL, Meny A, Aldhafri S, Banjar R, Alzahrani H. Efficacy of an acute bout of isometric wall squat exercise on pain sensitivity and clinical pain intensity in adults with knee osteoarthritis: a randomised controlled trial in outpatient physiotherapy clinics in Saudi Arabia. BMJ Open. 2025 Dec 11;15(12):e103756. doi: 10.1136/bmjopen-2025-103756. PMID 41381113